CLINICAL TRIAL: NCT02480452
Title: Brain Lesions in Relation to Motor Profiles of Children With Cerebral Visual Impairment.
Status: Completed | Type: Observational
Sponsor: Universitaire Ziekenhuizen KU Leuven (Other)
Responsible Party: Sponsor
Other Study IDs: S57844
Record Dates: First submitted 2015-06-21; First posted 2015-06-24 (Estimated); Last update posted 2023-01-27 (Actual); Status verified 2015-06

CONDITIONS: Visual Pathway Diseases; Neuroimaging

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- CVI: All children consulting at the CVI clinic (with suspicion of CVI) receiving a diagnosis of CVI
- no CVI: All children consulting at the CVI clinic (with suspicion of CVI) not receiving a diagnosis of CVI

SUMMARY:
The overall goal of this research proposal is the early prediction of the emergence of CVI and its characteristics on the basis of neuroimaging data.

The different steps that will be taken to achieve this goal will be:

1. To characterize CVI deficits in children;
2. To correlate the CVI characteristics with their motor profiles;
3. To characterize brain lesions in children with CVI;
4. To link the motor profile, CVI profile and brain metrics of the children.

Over the last 10 years, 488 children with and without CP have consulted at the CVI clinic in Leuven. All these children had a comprehensive visual perceptual assessment, cognitive evaluation and an ophthalmological assessment. Summarizing these data results in a quantitative visual perceptual profile for each individual patient. The goal is to prospectively extend this database to a number of 600 children. The project's primary objective is to relate the presence of CVI to the motor profiles of these children.

Of these 488 children, 300 have an MRI available. The goal is to analyze the retrospective MRI data of this clinical group and to prospectively extend this database by reassuring newly registered children will receive MRI with DTI. This will allow the investigation of the correlation between the brain metrics and the CVI characteristics in a large cohort.

DETAILED DESCRIPTION:
Objective 1 &2: to investigate the relationship between the presence of CVI and the motor profiles of children diagnosed with CVI.

Part 1 Retrospective data A database, registering all children diagnosed with or at risk for CVI, is available through the Centre For Developmental Disabilities, Leuven. All these children have consulted at the CVI clinic. Their developmental age ranges between 3 and 6 years. All these children have had a thorough work-up, so that information is available regarding the diagnosis of CVI (L94 visual perceptual battery test score10 and CVI questionnaire11), the cognitive abilities of the child (performance and verbal IQ using WISC-II, SON-R or WPPSI-III-NL) together with the test results regarding motor functioning: visuospatial functioning (VMI12 and TVPS13), motor coherence tasks and gross motor function (movement ABC14).

All children standardly received a complete ophthalmological assessment. The consensus eye protocol, as introduced by the Flemish working group on CVI, was performed in each child, evaluating fixation of eyes, position and motility, acuity, refraction, contrast sensitivity, visual field, visual attention and viewing distance.

Part 2 Prospective data The database will continuously be updated and therefore, data from all new consulting children will be added consecutively.

Prospectively, a new test for the diagnosis of CVI will be applied. It concerns a newly developed tool for diagnosis of CVI, based on the L-POST and developed in collaboration with the research group of J. Wagemans. Normative data have been gathered for the age ranges 3 to 6 years. The diagnosis of CVI is made by comparing the results of the visual perceptual tests to the developmental age of the child, with a result <Pc 5 necessary for CVI to be confirmed.15 These tests are standardly performed during the consultations and do not require any additional time nor tests.

As in the retrospective cohort, cognitive and motor assessments will be performed.

The retrospective and prospective data together will allow us to relate the CVI characteristics to the motor profiles of the children.

Objective 3&4: To build a prediction model based on the correlations found between brain metrics and CVI characteristics.

Part 1 Retrospective data If clinically mandatory, children had an MRI of the brain performed either around the time of their CVI diagnosis or earlier in case they had a pre-existing condition. We will correlate quantified CVI measures to the location and extent of the underlying brain lesions, if present, and the (lack of) white matter tract integrity using structural MRI and DTI. Our neuromotor research team (FABER-UZ Leuven, CP reference centre) already developed a specific standardized imaging protocol for CP, mainly directed at detection of white matter damage. This protocol includes at least FLAIR, MPRAGE, and DTI sequences. First of all, the qualitative classification of the SCPE will be used to classify conventional MRI.16 In children with dyskinetic CP, the classification of K. Himmelmann can additionally be performed.17 To perform a more comprehensive qualitative and semi-quantitative evaluation of brain lesions visible on conventional MRI, the FIORI classification scale, recently developed in collaboration with our group, will be used.18 Additionally, quantitative evaluations of microstructural brain lesions will be realized through the reconstruction of white matter tracts (e.g. inferior longitudinal fasciculus) using DTI. In this way, we will be able to link a set of neural parameters to measures of visual perceptual deficits. The goal of this study is to identify MRI- and DTI-parameters that are able to discriminate between children with and without CVI on the one hand and between different CVI patterns on the other hand. We expect that combinations and interactions of different MRI- and DTI-parameters, instead of single parameters, will be better suited for prognosis of the presence of CVI and of its characteristics. If possible, supplementary volumetric data will be gathered using the same scan.

Over the last 10 years, we have already collected a large dataset of children with and without CP, seen at the CVI clinic in Leuven. Of these 400 children, 300 have an MRI available. The diagnosis of CVI was made when results on the visual perceptual tests were at a level <Pc 5 for the developmental age. The retrospective MRI data of this clinical group will be thoroughly analyzed in the various ways described above and subsequently correlated to the visual perceptual data. In this way, we will obtain a clearer insight in the relation between metrics of brain lesions and CVI characteristics.

Part 2 Prospective data Prospective data will be gathered in a similar way as the retrospective data collection. Children will preferably receive an MRI with DTI around the age of 5 years. Around this age, with the help of a child-friendly scanning protocol (developed by PhD student Marjolein Verly), anaesthesia can be avoided. In all children demonstrating clinical relevant CVI features, an MRI with DTI will be performed. Subsequently, data will be analyzed in a similar way as the retrospective MRI data.

The first part of the study is designed as a retrospective cohort study. Data is collected from the standardized tests that are routinely performed during the CVI consultations. Trained staff members of the Centre for Developmental Disabilities performed the tests.

1. Background information:

   Information regarding the age, the birth history and the school system the child is enrolled in.
2. CVI diagnostic data:

   * Ophthalmological assessment
   * CVI Flemish questionnaire for parents is a standardized questionnaire, developed by the Flemish working group on CVI to give an overall idea of the visual functioning of the child.11
   * The L94 visual perceptual battery is an object recognition test, comprising 8 visual perceptual tasks for which normative data are available for children aged between 2,75 and 6,5 years. In 5 computer tasks, the child is asked to identify everyday objects and thus is tested for semantic and perceptual categorization.10
   * Motion coherence tasks: specific tests evaluating motion coherence, motion speed, biological motion and form from motion tasks will be performed as well.
3. Cognitive functioning is evaluated using standardized testing by means of the WISC-II, SON-R or WPPSI-III-NL respectively. The exact test is selected based on the age, the mental and physical capacities of the child.
4. Visuospatial functioning:

   * The Beery-Buktenica developmental test of Visual-Motor Integration (VMI)12 is widely used to assess visual perceptual abilities. The VMI consists of three subtests. First, in the copy task, the individual is asked to copy geometric forms, arranged in order of increasing difficulty. Second, the visual perception task uses the same geometric forms but now asks the subject to search a specific form in a series of similar forms. Third, in the Motor Coordination Task the subject is asked to copy these drawings in a frame. The copy task predominantly relies on visuomotor abilities.
   * The Test of Visual Perceptual skills (TVPS)13 is a motor-free task assessing different categories of visual perceptual skills: Visual Discrimination, Visual Memory Visual-Spatial Relations, Visual Form Consistence, Visual Sequential Memory, Visual Figure Ground and Visual Closure.
5. Motor functioning is evaluated using the Movement ABC-214, that contains 8 tasks for each age range in three areas: Manual Dexterity, Ball Skills and Static and Dynamic Balance. A profile of a child's performance over the different sections of the test can be examined. The assessment is paralleled by an observational approach with item-specific observations designed to help the examiner focus on the perceptual-motor aspects and overall evaluation to pinpoint emotional and motivational difficulties the child may have in relation to motor tasks. The Movement ABC-2 Checklist takes assessment into the everyday situations in which the child has to function. It provides an economical means of assessing groups of children through classroom assessment.
6. Neurological assessment: a standardized clinical examination is routinely performed to evaluate neurological signs such as abnormal muscle tone and pathological reflexes.
7. Brain imaging using structural MRI and DTI is evaluated using a specific standardized imaging protocol, mainly directed at detection of white matter damage.

The second part of the study is the prospective continuation of the retrospective cohort study. As during the retrospective part of the study, the same standardized tests are routinely performed during the CVI consultations and performed by the trained staff members of the Centre for Developmental Disabilities. However, prospectively, some additional tests will be performed

1. An assessment battery based on the L-POST15 will complement the diagnosis of the L94. The L-POST is a tool for visual perceptual assessment in adults. The subtests can be classified in 5 visual domains: (1) object recognition in a scene, (2) degraded object recognition , (3) motion perception, (4) global and local processing, and (5) visual memory. The test is computer based and does not require motor actions. Normative data are currently being gathered for the age ranges 3 to 6 years. The diagnosis of CVI is made by comparing the results of the visual perceptual tests to the developmental age of the child, with a result <Pc 5 necessary for CVI to be confirmed.15
2. The MRI and DTI will be performed whenever clinically relevant.

ELIGIBILITY:
Inclusion Criteria:

* mental age between 3 y and 6 y
* suspicion of CVI

Exclusion Criteria:

* mental age below 3y

Ages: 3 Years to 6 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: All children with a mental age between 3 and 6 years old consulting at the CVI clinic
Sampling Method: Non-Probability Sample
Enrollment: 600 (Estimated)
Dates: Start 2015-05; Primary Completion 2018-06 (Actual); Study Completion 2019-06 (Actual)

PRIMARY OUTCOMES:
L94 visual perceptual battery | baseline
  Diagnostic assessment for CVI
FIORI scale | baseline
  Outcome parameters for quantitative scoring of brain MRI

SECONDARY OUTCOMES:
Visual motor assessment | baseline
  Visual Motor Integration Test (VMI); Test of Visual Percepual Skills (TVPS)
Gross motor function | baseline
  Movement ABC
Motion coherence tasks | baseline
  Standardized test evaluating motion coherence

CONTACTS AND LOCATIONS:
Locations (1):
- Centre for Developmental disabilities, Leuven, Flanders, Belgium